CLINICAL TRIAL: NCT00508014
Title: Concurrent Peer Review Visits to Reduce Cardiovascular Risk Factors
Brief Title: Assessing the Effectiveness of Concurrent Peer Review for Patients With Cardiovascular Disease and Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Kevin Fiscella, Tenured Professor, University of Rochester
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 59768
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular disease; Diabetes; Quality improvement; Peer review
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): usual care
  Interventions: Other: Usual Care
- Concurrent Peer Review Visit (Experimental): See description of interventioin
  Interventions: Behavioral: Concurrent Peer Review visit

INTERVENTIONS:
Other: Usual Care — Usual Care with primary care provider during time period
  Arms: Control
Behavioral: Concurrent Peer Review visit — Participants are offered an office visit with a peer of their clinician primary clinician. This office visit is structured and focused on blood pressure, diabetic, and/or lipid control with decision support available at point of care
  Arms: Concurrent Peer Review Visit

SUMMARY:
We will assess the impact of concurrent peer review vists on blood pressure, cholesterol and diabetes control. Concurrent peer review (CPR) visits refer to special offic visits by patients to a clinician (physician, nurse practitioner, or physician assistant) other than than their primary care provider that are specifically designed to improve care for diabetes and cardiovascular disease.

DETAILED DESCRIPTION:
This project aims to reduce racial and ethnic disparities in health care by improving cardiovascular and diabetes management among poor and minority patients. We propose to implement and evaluate an innovative, but practical intervention: CPR visits. CPR visits are designed to minimize competing demands for clinicians and reduce clinical inertia by focusing clinician and patient attention on optimizing cardiovascular and/or diabetes management and disease control and through use of clinician prompts and decision support at the point of care. Following training of clinician staff, CPR visits will be implemented within two sites of a single community health center (Westside Health Services, Inc). Patients will be randomly assigned one CPR visit with a clinician other than their primary care clinician or to usual care. The primary study outcome will include control of hypertension, diabetes, and lipids. Secondary outcomes will include process measures for cardiovascular and diabetes care. Both personnel and data collection infrastructure will build on the existing Health Disparities Collaborative at Westside. A research team from the University of Rochester will assist in the implementation of study design. This team will lead both the quantitative and qualitative evaluation of the project including outcome and process measures. Project findings offer promise for improving care to underserved populations through dissemination and implementation of a feasible strategy among practices caring for the underserved. Findings will be disseminated nationally in conjunction with the Robert Wood Johnson Foundation, the National Association of Community Health Centers, and the National Health Disparities Collaborative and through publication in the peer reviewed literature and presentation at national conferences.

ELIGIBILITY:
Inclusion Criteria:

* Active patient at Westside Health Services.
* Currently enrolled in the Health Disparities Collaborative at WHS.
* At least one visit to primary care provider in past year.
* Any of the following documented during the preceding three months:
* BP not at goal e,g. (BP 140/80 or greater unless has DM, CAD or CRI then BP greater than 130/80), LDL-C not at goal (level dependent on absolute ATP III CVD risk) or glycated hemoglogin 7 percent or higher

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 727 (Actual)
Dates: Start 2006-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Mean change in blood pressure, glycated hemoglobin, and LDL-cholesterol between baseline and follow-up | 7 months

SECONDARY OUTCOMES:
Use of aspirin, ACE inhibiters/ARBs (diabetic patients), pneumonia vaccine updated, diabetic foot exam, diabetic microalbumuria check, retinal exam, smoking cessation counseling, dental visit, and self management goal | one year

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Fiscella, MD, MPH, Study Director — University of Rochester
Locations (1):
- Westside Health Services, Inc, Rochester, New York, United States

REFERENCES:
- See also: Robert Wood Johnson Foundation Website on Grantees — http://www.solvingdisparities.org/